CLINICAL TRIAL: NCT05090566
Title: A PHASE 1B/2, OPEN LABEL UMBRELLA STUDY OF ELRANATAMAB (PF-06863135), A B-CELL MATURATION ANTIGEN (BCMA) CD3 BISPECIFIC ANTIBODY, IN COMBINATION WITH OTHER ANTI-CANCER TREATMENTS IN PARTICIPANTS WITH MULTIPLE MYELOMA
Brief Title: MagnetisMM-4: Umbrella Study of Elranatamab (PF-06863135) in Combination With Anti-Cancer Treatments in Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071004; Umbrella Study (Other: Alias Study Number); MAGNETISMM-4 (Other: Alias Study Number); 2021-003885-11 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: PF-06863135, Multiple Myeloma, BCMA, elranatamab, bispecific antibody, MagnetisMM-4
MeSH Terms: conditions — Multiple Myeloma | interventions — nirogacestat; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub-Study A (Experimental): BCMA-CD3 bispecific antibody + gamma secretase inhibitor
  Interventions: Drug: Elranatamab + Nirogacestat
- Sub-Study B (Experimental): BCMA-CD3 bispecific antibody + immunomodulatory drug
  Interventions: Drug: Elranatamab + lenalidomide + dexamethasone

INTERVENTIONS:
Drug: Elranatamab + Nirogacestat — BCMA-CD3 bispecific antibody + gamma secretase inhibitor
  Other Names: PF-06863135, Ogsiveo
  Arms: Sub-Study A
Drug: Elranatamab + lenalidomide + dexamethasone — BCMA-CD3 bispecific antibody + immunomodulatory
  Other Names: PF-06863135; Revlimid
  Arms: Sub-Study B

SUMMARY:
The purpose of this study is to determine the Recommended Phase 2 Dose and clinical benefit of elranatamab in combination with other anti-cancer therapies in participants with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory multiple myeloma with at least 3 prior lines of therapy
* Refractory to at least one IMiD, one proteasome inhibitor, and one anti-CD38 antibody
* Measurable disease defined by at least one of the following:

  1. Serum M-protein >/= 0.5 g/dL by SPEP
  2. Urinary M-protein excretion >/= 200 mg/24 hours by UPEP
  3. Serum immunoglobulin FLC >/= 10 mg/dL (>/= 100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio
* ECOG performance status 0 -1
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade </= 1

Exclusion Criteria:

* Active plasma cell leukemia
* Amyloidosis
* Stem cell transplant with 12 weeks prior to enrollment, or active GVHD
* POEMS syndrome
* Any active uncontrolled bacterial, fungal, or viral infection
* Impaired cardiovascular function or clinically significant cardiovascular diseases within 6 months prior to enrollment
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of study treatment (whichever is longer)
* Sub-Study A Only: Previous treatment with BCMA bispecific antibody
* Sub-Study B Only: Previous treatment with BCMA directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Sub-Study A Phase 1: Dose Limiting Toxicity | approximately 35 days
  Number of participants with Dose Limiting Toxicity
Sub-Study A Phase 2: Objective Response Rate | assessed every 4 weeks (for approximately 2 years)
  Objective response rate (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Dose Limiting Toxicity | approximately 42 days
  Number of participants with Dose Limiting Toxicity

SECONDARY OUTCOMES:
Sub-Study A Phase 1: Objective Response Rate | assessed every 4 weeks (for approximately 2 years)
  Objective response rate (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Complete Response Rate | assessed every 4 weeks (for approximately 2 years)
  Complete response rate (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Time to Response | assessed every 4 weeks (for approximately 2 years)
  Time to response (IMWG criteria)
Sub-Study A Phase 1 and 2: Duration of Response | assessed every 4 weeks (for approximately 2 years)
  Duration of response (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Duration of Complete Response | assessed every 4 weeks (for approximately 2 years)
  Duration of complete response (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Progression Free Survival | assessed every 4 weeks (for approximately 2 years)
  Progression free survival (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Overall Survival | assessed for approximately 2 years
  Overall survival
Sub-Study A Phase 1 and Phase 2: Minimal Residual Disease Negativity Rate | assessed approximately every 12 months (for approximately 2 years)
  Minimal residual disease negativity rate (IMWG response criteria)
Sub-Study A Phase 1 and Phase 2: Frequency of Treatment-Emergent Adverse Events | assessed for approximately 2 years
  Type and severity per NCI CTCAE v5 (CRS and ICANS assessed per ASTCT criteria)
Sub-Study A Phase 1 and Phase 2: Frequency of Laboratory Abnormalities | assessed every cycle (each cycle approximately 28 days)
  Type and severity per NCI CTCAE v5
Sub-Study A Phase 1 and Phase 2: Immunogenicity of elranatamab in combination with nirogacestat | assessed approximately every 1 to 3 cycles (each cycle approximately 28 days)
  Anti-drug antibodies and neutralizing antibodies against elranatamab
Sub-Study A Phase 1 and Phase 2: Concentrations of elranatamab and/or nirogacestat | assessed approximately every 1 to 3 cycles (each cycle approximately 28 days)
  Pre-dose and post-dose concentrations of elranatamab; pre-dose concentrations of nirogacestat
Sub-Study A Phase 1: Maximum Observed Concentration (Cmax) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  Cmax for elranatamab administration
Sub-Study A Phase 1: Time to Maximum Concentration (Tmax) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  Tmax for elranatamab administration
Sub-Study A Phase 1: Area Under the Concentration versus Time Curve from Time 0 to the Last Measurable Concentration (AUClast) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  AUClast for elranatamab administration
Sub-Study B Phase 1 Escalation: Frequency of Treatment-Emergent Adverse Events | assessed for approximately 2 years
  Type and severity per NCI CTCAE v5 (CRS and ICANS assessed per ASTCT criteria)
Sub-Study B Phase 1 Escalation: Frequency of Laboratory Abnormalities | assessed every cycle (each cycle approximately 28 days)
  Type and severity per NCI CTCAE v5
Sub-Study B Phase 1 Escalation: Objective Response Rate | assessed every 4 weeks (for approximately 2 years)
  Objective response rate (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Complete Response Rate | assessed every 4 weeks (for approximately 2 years)
  Complete response rate (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Time to Response | assessed every 4 weeks (for approximately 2 years)
  Time to response (IMWG criteria)
Sub-Study B Phase 1 Escalation: Duration of Response | assessed every 4 weeks (for approximately 2 years)
  Duration of response (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Duration of Complete Response | assessed every 4 weeks (for approximately 2 years)
  Duration of complete response (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Progression Free Survival | assessed every 4 weeks (for approximately 2 years)
  Progression free survival (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Overall Survival | assessed for approximately 2 years
  Overall survival
Sub-Study B Phase 1 Escalation: Minimal Residual Disease Negativity Rate | assessed approximately every 12 months (for approximately 2 years)
  Minimal residual disease negativity ratio (IMWG response criteria)
Sub-Study B Phase 1 Escalation: Immunogenicity of elranatamab in combination with lenalidomide | assessed approximately every 1 to 3 cycles (each cycle approximately 28 days)
  Anti-drug antibodies and neutralizing antibodies against elranatamab
Sub-Study B Phase 1 Escalation: Concentrations of elranatamab and/or lenalidomide | assessed approximately every 1 to 3 cycles (each cycle approximately 28 days)
  Pre-dose and post-dose concentrations of elranatamab, pre-dose concentrations of lenalidomide
Sub-Study B Phase 1 Escalation: Maximum Observed Concentrations (Cmax) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  Cmax for elranatamab administration
Sub-Study B Phase 1 Escalation: Time to Maximum Concentration (Tmax) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  Tmax for elranatamab administration
Sub-Study B Phase 1 Escalation: Area Under the Concentration versus Time Curve from Time 0 to the Last Measurable Concentration (AUClast) for elranatamab | assessed after first elranatamab dose (approximately 3-7 days)
  AUClast for elranatamab administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (21):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner Gateway Medical Pavilion, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner Health d.b.a. Banner MD Anderson Cancer Center, Phoenix, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Clinical Research Advisors, Encino, California
  - Clinical Research Advisors, Los Angeles, California
  - Cedars Sinai Medical Center Oncology IDS Pharmacy Attn:Suwicha Limvorasak ,PharmaD, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute (SOCCI), Los Angeles, California
  - Cedars-Sinai Tarzana, Tarzana, California
  - Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami, Coral Gables, Florida
  - Sylvester Comprehensive Cancer Center- Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - UHealth Tower, Miami, Florida
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - OIDS, The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Also Imaging Facility), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Canada (3):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071004